CLINICAL TRIAL: NCT04241497
Title: Home-based Exercise Training in Patients With Pulmonary Arterial Hypertension: Effect on Skeletal Muscular Function and Metabolism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Marius Lebret, Post-doctoral fellow, Laval University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HTAP A DOM
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Pulmonary Arterial Hypertension; Exercise Training; Home-based Rehabilitation; Exercise Capacity; Muscle Metabolism; Muscle Function; Lipid Infiltration; Oxidative Metabolism
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Pulmonary Arterial Hypertension (Experimental): 12 weeks home-based rehabilitation
  Interventions: Behavioral: Home-based rehabilitation

INTERVENTIONS:
Behavioral: Home-based rehabilitation — 1 supervised exercise session at the hospital; 3 weeks of supervised home-based exercise training (3x/week); 9 weeks of unsupervised home-based exercise training (3x/week)

SUMMARY:
Pulmonary Arterial Hypertension has gone from a disease that causes rapid death to a more chronic condition. Yet, improved survival is associated with major challenges for clinicians as most patients remain with poor quality of life and limited exercise capacity. The effects of exercise training on exercise capacity have been largely evaluated and showed an improvement in 6-minutes walking distance (6MWD), peak V'O2. It is also known that exercise program improves quality of life. Maximal volitional and nonvolitional strength of the quadriceps are reduced in patients with Pulmonary Arterial Hypertension and correlated to exercise capacity. Moreover, on the cellular level, alterations are observed in both the respiratory as well as the peripheral muscles. Muscle fiber size has been reported to be decreased in some studies or conversely unaltered in human and animal models. Reduction in type I fibers and a more anaerobic energy metabolism has also been reported, but not in all studies. Likewise, a loss in capillary density in quadriceps of patients with Pulmonary Arterial Hypertension and rats has been reported, but could not be confirmed in other studies. While the impact of exercise training on clinical outcomes such as exercise capacity or quality of life is well known, this data highlight the fact that the underlying causes of peripheral muscle weakness as well as the mechanisms underlying the clinical improvements observed with exercise programs are not completely understood. Improvement of muscle cell metabolism in part via the enhancement of oxidative cellular metabolism and decrease in intracellular lipid accumulation may play a role in improving muscle function and exercise capacity.

In this study, we intend to evaluate the impact of a 12 weeks home-based rehabilitation program on peripheral muscle function and metabolism, focusing on lipid infiltration, oxidative metabolism and epigenetic factors that can be involved in metabolic syndrome, in patients with Pulmonary Arterial Hypertension.

DETAILED DESCRIPTION:
The 12 weeks home-based rehabilitation program is detailed as follows:

* 1st sessions at the hospital, in the presence of a physiotherapist/kinesiologist
* 3 weeks of supervised home-based rehabilitation (using a telemonitoring system) 3 times a weeks
* 9 weeks of unsupervised home-based rehabilitation (one phone call a week)

Patients will be evaluated at baseline and at endpoint (12 weeks)

ELIGIBILITY:
Inclusion Criteria:

* Men or women > 18 years old
* Pulmonary Arterial Hypertension group 1: idiopathic, genetics, drug or toxin-induced, associated with connective tissue, HIV, portal hypertension, congenital heart disease.
* Diagnosis performed by right heart catheterization with Pulmonary Arterial Pressure⩾ 20 mmHg, pulmonary artery occlusion pressure <15 and pulmonary vascular resistance >3 Wood units
* New York Heart Association II or III and a 6-Minute Walk Test < 500m
* Patient stable without therapeutic modification within the last 3 months
* Patient having wireless internet at home
* Consciously informed and written by the patient

Exclusion Criteria:

* Syncope within the last 6 month
* Metabolic comorbidity (eg Diabetes)
* Musculoskeletal impairment that does not allow physical exercise
* Patient unable or with contraindications to perform a cardio pulmonary exercise testing
* Patient with pulmonary veno-occlusive disease
* Presence of a permanent pacemaker or other contraindication to MRI
* Pregnant or breastfeeding woman
* Age <18 years

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Epigenetic factors influencing muscle metabolism | Changes between baseline and 12 weeks of exercise rehabilitation
  Transcriptome analysis using RNA-seq

SECONDARY OUTCOMES:
Intramyocellular lipid accumulation | Changes between baseline and 12 weeks of exercise rehabilitation
  H-magnetic resonance spectroscopy and Oil red O technique
Muscular mitochondrial phosphorylation (ATP synthesis) | Changes between baseline and 12 weeks of exercise rehabilitation
  phosphorus-31 Magnetic resonance spectroscopy saturation transfer
Proportion of muscle fiber types | Changes between baseline and 12 weeks of exercise rehabilitation
  Ethanol modified technique
HbA1c | Changes between baseline and 12 weeks of exercise rehabilitation
  Serum HbA1c
Insulin | Changes between baseline and 12 weeks of exercise rehabilitation
  Serum Insulin
Glucose | Changes between baseline and 12 weeks of exercise rehabilitation
  Serum glucose
Apolipoprotein A1 | Changes between baseline and 12 weeks of exercise rehabilitation
  Serum Apolipoprotein A1
Adiponectin | Changes between baseline and 12 weeks of exercise rehabilitation
  Serum Adiponectin
Leptin | Changes between baseline and 12 weeks of exercise rehabilitation
  Serum leptin
Volitional strength quadriceps | Changes between baseline and 12 weeks of exercise rehabilitation
  Maximal Voluntary force using isometric force meter
Non-volitional strength of the quadriceps | Changes between baseline and 12 weeks of exercise rehabilitation
  Maximal non-Voluntary force using isometric force meter and magnetic stimulation of the femoral neve
Maximal exercise capacity | Changes between baseline and 12 weeks of exercise rehabilitation
  Cardio-pulmonary exercise testing on a cycloergometer
Functional Exercise capacity | Changes between baseline and 12 weeks of exercise rehabilitation
  6-MWD
Quality of life (QOL) | Changes between baseline and 12 weeks of exercise rehabilitation
  Cambridge Pulmonary Hypertension Outcome Review (CAMPHOR) questionnaire. The CAMPHOR questionnaire contains 65 items in total, 25 relating to symptoms, 15 relating to activities, and 25 relating to QoL. It is negatively weighted; a higher score indicates worse QoL and greater functional limitation. Symptom and QoL items are both scored out of 25: "yes/true" scores 1 and "no/not true" scores 0. Activity items have three possible responses (score 0-2), giving a score out of 30. Each CAMPHOR assessment takes an average of 10 min

CONTACTS AND LOCATIONS:
Locations (1):
- University Institute of Cardiology and Respirology of Quebec, Québec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Grunig E, Lichtblau M, Ehlken N, Ghofrani HA, Reichenberger F, Staehler G, Halank M, Fischer C, Seyfarth HJ, Klose H, Meyer A, Sorichter S, Wilkens H, Rosenkranz S, Opitz C, Leuchte H, Karger G, Speich R, Nagel C. Safety and efficacy of exercise training in various forms of pulmonary hypertension. Eur Respir J. 2012 Jul;40(1):84-92. doi: 10.1183/09031936.00123711. Epub 2012 Feb 9. PMID 22323570
- [Result] Ehlken N, Lichtblau M, Klose H, Weidenhammer J, Fischer C, Nechwatal R, Uiker S, Halank M, Olsson K, Seeger W, Gall H, Rosenkranz S, Wilkens H, Mertens D, Seyfarth HJ, Opitz C, Ulrich S, Egenlauf B, Grunig E. Exercise training improves peak oxygen consumption and haemodynamics in patients with severe pulmonary arterial hypertension and inoperable chronic thrombo-embolic pulmonary hypertension: a prospective, randomized, controlled trial. Eur Heart J. 2016 Jan 1;37(1):35-44. doi: 10.1093/eurheartj/ehv337. Epub 2015 Jul 31. PMID 26231884
- [Result] Grunig E, Eichstaedt C, Barbera JA, Benjamin N, Blanco I, Bossone E, Cittadini A, Coghlan G, Corris P, D'Alto M, D'Andrea A, Delcroix M, de Man F, Gaine S, Ghio S, Gibbs S, Gumbiene L, Howard LS, Johnson M, Jureviciene E, Kiely DG, Kovacs G, MacKenzie A, Marra AM, McCaffrey N, McCaughey P, Naeije R, Olschewski H, Pepke-Zaba J, Reis A, Santos M, Saxer S, Tulloh RM, Ulrich S, Vonk Noordegraaf A, Peacock AJ. ERS statement on exercise training and rehabilitation in patients with severe chronic pulmonary hypertension. Eur Respir J. 2019 Feb 28;53(2):1800332. doi: 10.1183/13993003.00332-2018. Print 2019 Feb. PMID 30578391
- [Result] Potus F, Malenfant S, Graydon C, Mainguy V, Tremblay E, Breuils-Bonnet S, Ribeiro F, Porlier A, Maltais F, Bonnet S, Provencher S. Impaired angiogenesis and peripheral muscle microcirculation loss contribute to exercise intolerance in pulmonary arterial hypertension. Am J Respir Crit Care Med. 2014 Aug 1;190(3):318-28. doi: 10.1164/rccm.201402-0383OC. PMID 24977625
- [Result] Malenfant S, Brassard P, Paquette M, Le Blanc O, Chouinard A, Nadeau V, Allan PD, Tzeng YC, Simard S, Bonnet S, Provencher S. Compromised Cerebrovascular Regulation and Cerebral Oxygenation in Pulmonary Arterial Hypertension. J Am Heart Assoc. 2017 Oct 12;6(10):e006126. doi: 10.1161/JAHA.117.006126. PMID 29025748
- [Result] Malenfant S, Potus F, Fournier F, Breuils-Bonnet S, Pflieger A, Bourassa S, Tremblay E, Nehme B, Droit A, Bonnet S, Provencher S. Skeletal muscle proteomic signature and metabolic impairment in pulmonary hypertension. J Mol Med (Berl). 2015 May;93(5):573-84. doi: 10.1007/s00109-014-1244-0. Epub 2014 Dec 30. PMID 25548805